CLINICAL TRIAL: NCT05991921
Title: The Effect of TENS Applied in the Early Postpartum Period on Incision Healing, Pain and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assit. Prof, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023/ 02- 13
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Recovery; Wound Healing; Postpartum Comfort; Postpartum Pain
Keywords: Transcutaneous Electrical Nerve Stimulation; wound healing; cesarean section; pain; comfort; Recovery; postpartum period
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study was designed as randomized, single-blind, placebo-controlled.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Based on simple randomization, women were assigned to one of three groups: TENS (n=46), placebo (n=46), or control (n=46). For randomization, researcher 1 used the random number generation method available on the random.org site. These processes are hidden from the rest of the study. While TENS application in the research was carried out by researcher 1; It was conducted by researcher 2, who evaluated the participants for inclusion and exclusion criteria and collected the data, who did not know the distribution of the participants. Because sham device TENS was not applied to the control group, the participants were able to realize that they were assigned to the control group. Therefore, this study was considered a single-blind study. To provide blinding in the placebo group, the participants were hooked up to the TENS unit in exactly the same way as the participants in the TENS group. The active indicator of the unit emitted light and sound, but did not transmit electrical stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcutaneous Electrical Nerve Stimulation" (Experimental): TENS application, postpartum 10-12. at hours and 14-16. It was applied twice for 30 minutes each.Two pairs of TENS electrodes were placed on the upper and lower border of the cesarean section incision line. A total of 4 electrodes were used in a sterile package for each participant. TENS stimulation was applied at a frequency of 100 Hz and was increased starting from 0 mA. The participant's stimulation was fixed at the mA level, where he felt optimal but did not feel discomfort. All participants in the TENS, received all other routine obstetric care provided by hospital healthcare professionals.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation (TENS)
- Plasebo (Sham Comparator): Participants in the placebo group 10-12 postpartum. at hours and 14-16. Two pairs of TENS electrodes were placed at the same time as the intervention group. TENS electrodes were attached to the participants in this group for 30 minutes, the device was operated but no electric current was applied.
  Interventions: Other: Plasebo-Fake TENS
- Control (No Intervention): Participants in the control group were not dependent on TENS. All participants in the control group received all other routine obstetric care provided by hospital healthcare professionals.

INTERVENTIONS:
Other: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS application, postpartum 10-12. at hours and 14-16. It was applied twice for 30 minutes each. Researcher 1 programmed the TENS unit and was the only researcher who knew whether TENS was active or in placebo mode.
  Two pairs of TENS electrodes were placed on the upper and lower border of the cesarean section incision line. A total of 4 electrodes were used in a sterile package for each participant. TENS stimulation was applied at a frequency of 100 Hz and was increased starting from 0 mA. The participant's stimulation was fixed at the mA level, where he felt optimal but did not feel discomfort.
  The pretest data were applied to the participants who met the inclusion criteria and volunteered to participate in the study, by the researcher 2 in the patient rooms 10 hours after the cesarean section. Post-test data were obtained by the same investigator 16 hours after cesarean section.
  Arms: Transcutaneous Electrical Nerve Stimulation"
Other: Plasebo-Fake TENS — Participants in the placebo group 10-12 postpartum. at hours and 14-16. Two pairs of TENS electrodes were placed at the same time as the intervention group. TENS electrodes were attached to the participants in this group for 30 minutes, the device was operated but no electric current was applied.
  Arms: Plasebo

SUMMARY:
Objective: In this study, it was aimed to determine the effect of TENS applied in the early postpartum period after cesarean section on incision healing, pain and comfort.

Methods: This study was designed as randomized, single-blind, placebo-controlled. All participants signed an informed consent statement before starting the study. The study sample of 138 (TENS group n=46, placebo group n=46, control group n=46).

TENS application, postpartum 10-12. at hours and 14-16. It was applied twice for 30 minutes each. Researcher 1 programmed the TENS unit and was the only researcher who knew whether TENS was active or in placebo mode. The pretest data were applied to the participants who met the inclusion criteria and volunteered to participate in the study, in the patient rooms 10 hours after the cesarean section. Post-test data were obtained by the same investigator 16 hours after cesarean section. Data were obtained with Personal Information Form, Postoperative Recovery Index (PoRI), REEDA Scale, Visual Analogue Scale (VAS), and Postpartum Comfort Scale (PPCQ).

DETAILED DESCRIPTION:
Introduction The postpartum period is a period with biopsychosocial effects in the life of the mother and her family. The mode of delivery may affect the adaptation of the mother to the postpartum period. Most women can have a vaginal birth with professional support. However, vaginal delivery can be risky in cases of fetal distress, large fetus, head and pelvis incompatibility, fetal posture disorders, and maternal illness that may prevent vaginal delivery. In these cases, cesarean section is an important decision for the health of both mother and baby. However, cerzerian surgery also brings some risks. Pain in the short term, difficulty in the recovery of the mother, delayed mobilization, infection, exposure to a surgical operation and a decrease in maternal comfort due to these may cause many problems such as breastfeeding problems, decreased mother-baby bonding.

The presence of persistent pain after cesarean section is the result of post-operative inflammatory reactions and adversely affects the mother. In a study, it was reported that 75% of women experienced moderate or severe pain after cesarean section, and this pain was high in the first 24 hours. The duration of pain may be prolonged depending on the individual's perception of pain and response to pain. It delays early mobilization by delaying pain relief and reduces maternal comfort. Effective treatment of pain is very important economically and because of its unpleasant physiological and psychological consequences for the patient. Recently, many methods have been developed with pharmacological and non-pharmacological approaches to pain in women with severe pain after cesarean section, and it has been reported that they accelerate pain, maternal satisfaction, recovery time and delay the use of analgesics. These include TENS, acupuncture, breathing exercises, and psychotherapy.

Transcutaneous Electrical Nerve Stimulation (TENS) is a non-pharmacological, low-frequency electrotherapy technique. The mechanism of action of TENS is still unknown. It was first used in obstetrics in 1970. It has been reported in the literature that TENS is used in chronic pain such as post-operative pain, vaginal delivery pain, dysmenorrhea, angina pectoris, orofacial pain, dental procedures, physical trauma-broken ribs and minor medical procedures, low back pain. Despite the widespread use of TENS in vaginal labor pain, it has been included in systematic reviews for which evidence of benefit is insufficient. In addition, it has been reported that TENS is effective in wound healing and faster wound area reduction in some dermatological studies and plastic surgery. It has been reported that TENS supports the long-term retention of flaps and grafts after plastic surgery, thereby accelerating postoperative recovery and reducing necrosis. The effectiveness of TENS in wound healing has been associated with an increase in blood flow (Visconti et al., 2020). However, there is no study in the literature that determines the effect of TENS on incision healing, pain and comfort after cesarean section.

Considering the cesarean section rates in the world and in Turkey, the importance of these risks emerges. While the Dominican Republic ranks first with 56.4% in the WHO's cesarean section rates, Turkey ranks fourth in this ranking. The rate of cesarean section in Turkey was determined to be 52% in 2018, according to the report of the Turkey Demographic and Health Survey (TNSA).

Considering the problems mentioned above, it is important to search for non-pharmacological interventions that will minimize health risks along with full holistic care for mothers in the post-cesarean period. Therefore, in this study, it was aimed to determine the effect of TENS applied in the early postpartum period at the end of the cesarean section on incision healing, pain and comfort.

Research questions:

1. TENS applied in the early postpartum period reduces the level of pain.
2. TENS applied in the early postpartum period improves incision healing and comfort

Materials and methods Study design This study was designed as randomized, single-blind, placebo-controlled. Study procedures were approved by the Inonu University Scientific Research and Publication Ethics Committee (Decision No: 2023/ 02-13), and comply with the ethical guidelines set forth in the Declaration of Helsinki. It was also conducted in accordance with Good Clinical Practice guidelines. All participants signed an informed consent statement before starting the study.

The study was conducted with women who gave birth by cesarean section in a hospital in eastern Turkey between January and August. Postoperative hospital stay for women is 48 hours postpartum, according to the policy of the Ministry of Health. Post cesarean section analgesia protocol is the same for all women in the hospital, except that analgesia is not applied. The routine analgesia protocol applied in the hospital is as follows: the first dose is administration of non-steroidal anti-inflammatory drugs (NSAIDS) within the first 30 minutes after surgery and then every 8 hours. Spinal anesthesia technique was used in all cesarean deliveries in the hospital.

Priori-power analysis was performed using the G*Power 3.1.9.2 program to calculate the appropriate sample size. The sample size of the study was calculated as at least 46 with an effect size of 0.40, a power of 0.95, and a margin of error of 0.05. These assumptions generated a sample size of 138 subjects, 46 per group (TENS group n=46, placebo group n=46, control group n=46).

Inclusion criteria for the study were as follows: (1) 18 years of age or older, (2) having a single healthy newborn. Exclusion criteria are as follows: (1) cesarean section under general anesthesia, (2) any postpartum complication (such as bleeding, hypertension), (3) skin damage at TENS application sites, (4) morbidly obese, (5) cardiac women using a pacemaker or automated implanted cardiac defibrillator, (6) previously using TENS, (7) receiving repeated doses of analgesics other than those routinely administered after surgery.

Randomization and blinding Based on simple randomization, women were assigned to one of three groups: TENS (n=46), placebo (n=46), or control (n=46). For randomization, researcher 1 used the random number generation method available on the random.org site. These processes are hidden from the rest of the study. While TENS application in the research was carried out by researcher 1; It was conducted by researcher 2, who evaluated the participants for inclusion and exclusion criteria and collected the data, who did not know the distribution of the participants. Because sham device TENS was not applied to the control group, the participants were able to realize that they were assigned to the control group. Therefore, this study was considered a single-blind study. To provide blinding in the placebo group, the participants were hooked up to the TENS unit in exactly the same way as the participants in the TENS group. The active indicator of the unit emitted light and sound, but did not transmit electrical stimulation.

Interventions TENS application, postpartum 10-12. at hours and 14-16. It was applied twice for 30 minutes each. Researcher 1 programmed the TENS unit and was the only researcher who knew whether TENS was active or in placebo mode.

Two pairs of TENS electrodes were placed on the upper and lower border of the cesarean section incision line. A total of 4 electrodes were used in a sterile package for each participant. TENS stimulation was applied at a frequency of 100 Hz and was increased starting from 0 mA. The participant's stimulation was fixed at the mA level, where he felt optimal but did not feel discomfort.

Participants in the placebo group 10-12 postpartum. at hours and 14-16. Two pairs of TENS electrodes were placed at the same time as the intervention group. TENS electrodes were attached to the participants in this group for 30 minutes, the device was operated but no electric current was applied. Participants in the control group were not dependent on TENS. All participants in the TENS, placebo, and control group received all other routine obstetric care provided by hospital healthcare professionals.

Data collection The pretest data were applied to the participants who met the inclusion criteria and volunteered to participate in the study, by the researcher 2 in the patient rooms 10 hours after the cesarean section. Post-test data were obtained by the same investigator 16 hours after cesarean section. Data were obtained with Personal Information Form, Postoperative Recovery Index (PoRI), REEDA Scale, Visual Analogue Scale (VAS), and Postpartum Comfort Scale (PPCQ). Data collection was carried out by researcher 2. The researcher received consent from 2 participants and administered a pre-test to the participants who agreed to participate in the study. After the pretest data were completed, researcher 1 performed the first TENS application. After researcher 1 completed the second TENS application, researcher 2 collected post-test data. Researchers entered the patient rooms separately. These processes were not shared with other participants in the study.

The Personal Information Form includes the descriptive characteristics of the participants such as age, education level, employment status, income level and number of births.

The PoRI index consists of 5 sub-dimensions and 25 items. Sub dimensions; psychological symptoms, physical activities, appetite symptoms, intestinal symptoms, and general symptoms. The scores of the items in the sub-dimensions are summed, their averages are calculated, and the sub-dimension scores are determined. For the PoRI total score, all 25 items are summed and averaged. High scores obtained from the index indicate that there are more problems in postoperative recovery, while low scores indicate that recovery is easier after surgery.

The REEDA scale is used to evaluate cesarean section incision wounds. This scale covers five factors that indicate wound healing: redness, edema, echymosis, discharge and approximation. Each of the improvement factors is evaluated by giving 0, 1, 2 and 3 points. The sum of the scores obtained as a result of the evaluation of the five categories forms the REEDA score. The lowest score is 0, the highest score is 15. Lower scores represent better wound healing. REEDA is a standardized scale with proven reliability and validity. The investigators chose to use the REEDA scale in this study, as it has been shown to be valid for the measurement of wound healing after Serzerian.

VAS was used to assess incision site pain severity. VAS is a scale created in the range of 0-100 mm. According to the scale, a score of 0 mm indicates that the pain is not severe at all, and a score of 100 mm indicates that the pain is very severe.

The PPCQ was developed to measure the level of postpartum comfort. The scale consists of 3 sub-dimensions and 34 items. Sub dimensions; physical comfort (components related to physical and bodily perceptions), psychospiritual comfort (components related to spiritual and psychology), sociocultural comfort (components related to interpersonal, family and social relations, finance and support systems). The total score of the scale ranges from 34 to 170. The increase in the average score obtained from the total and sub-dimension averages of the scale indicates that the comfort level also increases.

Statistical analysis Statistical calculations were made using IMB SPSS version 25.0 for Windows. Qualitative variables were presented as frequency and percentage, and quantitative variables as mean ± standard deviation. The descriptive characteristics of the participants were compared with the chi-square test. Paired-samples t-test was used for in-group comparisons and one-way analysis of variance (ANOVA) was used for inter-group comparisons to test the intervention effects, since the condition of normal distribution was met. When the difference between groups was significant, post-hoc multiple comparison was analyzed with Tukey's test.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* having a single healthy newborn.

Exclusion Criteria:

* cesarean section under general anesthesia,
* any postpartum complication (such as bleeding, hypertension),
* skin damage at TENS application sites,
* morbidly obese,
* cardiac women using a pacemaker or automated implanted cardiac defibrillator,
* previously using TENS,
* receiving repeated doses of analgesics other than those routinely administered after surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — being ≥18 years old
Enrollment: 138 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
Postoperative Recovery Index (PoRI) | Change from PoRI at 16 hours after cesarean section
  The PoRI index consists of 5 sub-dimensions and 25 items. Sub dimensions; psychological symptoms, physical activities, appetite symptoms, intestinal symptoms, and general symptoms. The scores of the items in the sub-dimensions are summed, their averages are calculated, and the sub-dimension scores are determined. For the PoRI total score, all 25 items are summed and averaged. High scores obtained from the index indicate that there are more problems in postoperative recovery, while low scores indicate that recovery is easier after surgery.

SECONDARY OUTCOMES:
REEDA Scale | Change from REEDA at 16 hours after cesarean section
  The REEDA scale is used to evaluate cesarean section incision wounds. This scale covers five factors that indicate wound healing: redness, edema, echymosis, discharge and approximation. Each of the improvement factors is evaluated by giving 0, 1, 2 and 3 points. The sum of the scores obtained as a result of the evaluation of the five categories forms the REEDA score. The lowest score is 0, the highest score is 15. Lower scores represent better wound healing. REEDA is a standardized scale with proven reliability and validity. We chose to use the REEDA scale in this study, as it has been shown to be valid for the measurement of wound healing after Serzerian.

OTHER OUTCOMES:
Visual Analogue Scale (VAS) | Change from REEDA at 16 hours after cesarean section
  VAS was used to assess incision site pain severity. VAS is a scale created in the range of 0-100 mm. According to the scale, a score of 0 mm indicates that the pain is not severe at all, and a score of 100 mm indicates that the pain is very severe.
Postpartum Comfort Scale (PPCQ) | Change from REEDA at 16 hours after cesarean section
  The PPCQ was developed to measure the level of postpartum comfort. The scale consists of 3 sub-dimensions and 34 items. Sub dimensions; physical comfort (components related to physical and bodily perceptions), psychospiritual comfort (components related to spiritual and psychology), sociocultural comfort (components related to interpersonal, family and social relations, finance and support systems). The total score of the scale ranges from 34 to 170. The increase in the average score obtained from the total and sub-dimension averages of the scale indicates that the comfort level also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabanci Baransel E, Barut S, Ucar T. The Effects of Transcutaneous Electrical Nerve Stimulation Applied in the Early Postpartum Period After Cesarean Birth on Healing, Pain, and Comfort. J Midwifery Womens Health. 2024 Sep-Oct;69(5):681-688. doi: 10.1111/jmwh.13625. Epub 2024 Mar 12. PMID 38470299